CLINICAL TRIAL: NCT04056377
Title: The Exercise, Arterial Modulation and Nutrition in Youth South Africa (ExAMIN Youth SA) Study
Brief Title: Exercise, Arterial Modulation and Nutrition in Youth South Africa Study
Acronym: ExAMIN-Youth
Status: Active, not recruiting | Type: Observational
Sponsor: North-West University, South Africa (Other)
Collaborators: National Research Foundation of South Africa (Other); Medical Research Council, South Africa (Other)
Responsible Party: Principal Investigator, Ruan Kruger, Professor, North-West University, South Africa
Other Study IDs: NWU-00091-16-A1
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Hypertension; Retinal Artery Stenosis; Childhood Obesity
Keywords: Hypertension; Retinopathy; Obesity; Arterial stiffness; Physical inactivity
MeSH Terms: conditions — Hypertension; Pediatric Obesity; Retinal Diseases; Obesity; Sedentary Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biological samples for biomarker analyses (spot urine and saliva) were taken at baseline and also for each follow-up. Samples are preserved for both short and long-term at -80°C. We aim to assess a variety of traditional and new biomarkers related to hypertension and cardiovascular disease.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Black boys: 240 black boys were included in the study (mean age 7.5 years)
- Black girls: 339 black girls were included in the study (mean age 7.5 years)
- White boys: 239 white boys were included in the study (mean age 7.4 years)
- White girls: 224 white girls were included in the study (mean age 7.4 years)

SUMMARY:
The ExAMIN Youth SA study aims to generate new knowledge on the pathophysiology involved in early vascular aging among South African children and to identify early novel biological markers for predicting the subclinical development of hypertension and target organ damage related to cardiovascular disease. This study further implements state-of-the-art biochemical technology to measure a variety of biological markers including multiplex analyses and metabolomics. With the increasing prevalence of childhood hypertension and obesity, this study will be able to address especially behavioural contributors to hypertension development and to subsequently provide a backdrop for school-based primary prevention interventions.

DETAILED DESCRIPTION:
Background: The current global widespread incidence of obesity and early cardiovascular deterioration are two of the most important future health care challenges. Physical inactivity and its associated unhealthy dietary intake among adolescents are of great concern, especially in a South African setting in which no current monitoring occurs to describe the impact of this sedentary and unhealthy lifestyle on cardiovascular health. With the estimated global prevalence of elevated blood pressure among children between 12-25%, there is a definite need to contribute to the lack of population level data in South Africa and how lifestyle behaviours impact on the burden of non-communicable disease.

Main aim: Our current study aims to build on previous findings to identify potential contributing factors that may adversely affect health outcomes in South African children. Additionally, we will cross-compare data with international centres on these health outcomes, and finally develop predictive models on target organ damage at 4-years follow-up from baseline data.

Design/Methods: We phenotyped a cohort of 1065 primary school children (all sexes, all ethnic groups and ages 5-9 years) according to their physical fitness and coordination, their dietary behaviours, psychosocial behaviour and current cardiovascular state. Parents of participating children provided information on socio-demographics including data on education, employment, types of dwelling, household amenities and parents' marital status, health habits, and lifestyle. The children will underwent the following measurements: anthropometric measurements of height, weight, waist circumference, triceps and subscapular skinfolds; stable isotope and bioelectric impedance analysis to measure body composition; blood pressure along with pulse wave analysis and aortic pulse wave velocity, static retinal vessel analysis (without mydriasis); accelerometry and a standardised physical activity questionnaire to measure physical activity. Physical fitness measures included motor skills, coordination, flexibility and cardio-respiratory fitness. Urinalysis will include creatinine, albumin, electrolytes, nitrates, nitrites, dimethylarginines, malondialdehyde, glucose, cardiovascular and kidney multiplex panels, and targeted metabolomics. Salivary analyses will include sex hormones and cortisol.

Outcomes: The primary outcomes for the baseline analysis include blood pressure, pulse wave velocity and retinal vascular calibres to address micro- and macrovascular compromise in relation to behavioural risk factors. In the follow-up phase of the study we will include carotid intima media thickness and left ventricular mass as outcomes of baseline predictors.

Timetable: The project was approved and is endorsed by the District Director of the Department of Education, and was approved by the Health Research Ethics Committee of the North-West University on 10 may 2017 (NWU-00091-16-A1). Data collection started in September 2017 and baseline measurements were concluded on 30 April 2019. Follow-up assessments will commence immediately in subsequent years for the 4-year follow-up phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Children between ages 5 and 9 years (both sexes and all ethnicities).

Exclusion Criteria:

* Children who do not wish to participate or where the parents or caregivers did not provide permission.

Ages: 62 Months to 129 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population included 1103 children (at baseline) attending public primary schools in the Dr Kenneth Kaunda district, North West province, South Africa aged between 5 and 9 years of age. However, with a few missing (n=38) values of basic variables of interest such as sex, ethnicity or date of birth, we included a total 1065 children (mean age=7.44 years or 89.3 months). The majority of the participants were of African (n=579) and white (n=463) ethnicity, whereas only 2.2% (n=23) participants were of either Indian or mixed race. The sex distribution was similar in the white group, whereas the study unintentionally included more girls (58.5%) than boys (41.5%) in the black group.
Sampling Method: Non-Probability Sample
Enrollment: 1065 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine blood pressure classification among primary school children in South Africa | Through study completion, an average of 1 year
  Elevated blood pressure and stage 1 hypertension according to the American Academy of Pediatrics Clinical Practice Guidelines 2017 stratified for age, sex, weight and height. Automated oscillometric calculations of central systolic blood pressure and pulse wave velocity.
To determine overweight and obesity prevalence among primary school children in South Africa | Through study completion, an average of 1 year
  Overweight and obesity classification according to the World Health Organisation percentiles for childhood obesity
To identify novel biomarkers in predicting elevated blood pressure in primary school children from South Africa | Through study completion, an average of 1 year
  Multiplex analysis of cardiovascular and kidney related biomarkers, and subsequently metabolomics and hormone concentrations

SECONDARY OUTCOMES:
Associations of central blood pressure and aortic stiffness with physical fitness | Through study completion, an average of 1 year
  Physical fitness (cardiorespiratory fitness, coordination, endurance, speed, balance) and activity (accelerometry)
Associations of central blood pressure and aortic stiffness with body composition | Through study completion, an average of 1 year
  Anthropometry including body heigh, body weight, waist-to-height ratio, and body fat percentage
Associations of central blood pressure and aortic stiffness and dietary intake | Through study completion, an average of 1 year
  Healthy and unhealthy food consumption frequencies determined by validate survey to depict unhealthy and healthy food group patterns
Associations of central blood pressure and aortic stiffness and childhood adversity | Through study completion, an average of 1 year
  Early life stress events as quantified by validated psychosocial questionnaires.

OTHER OUTCOMES:
Determine the change in blood pressure over a 4-year follow-up period in primary school children of South Africa | Through study completion, 4 years after baseline measurements
  Automated oscillometric calculations of central systolic blood pressure and pulse wave velocity at baseline and 4-years follow-up
Determine baseline predictors of target organ damage markers after a 4-year follow-up period in primary school children of South Africa | Through study completion, 4 years after baseline measurements
  Target organ damage will be assessed at follow-up by carotid intima media thickness and left ventricular mass.

CONTACTS AND LOCATIONS:
Locations (1):
- Hypertension in Africa Research Team (HART), North-West University, Potchefstroom, North West, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kochli S, Smith W, Lona G, Goikoetxea-Sotelo G, Breet Y, Botha-Le Roux S, Mokwatsi GG, Kruger R, Hanssen H. Obesity, blood pressure and retinal microvascular phenotype in a bi-ethnic cohort of young children. Atherosclerosis. 2022 Jun;350:51-57. doi: 10.1016/j.atherosclerosis.2022.04.018. Epub 2022 Apr 21. PMID 35490596
- [Derived] Kruger R, Kruger HS, Monyeki MA, Pienaar AE, Roux SB, Gafane-Matemane LF, Smith W, Mels CMC, Lammertyn L, Brits JS, Hanssen H. A demographic approach to assess elevated blood pressure and obesity in prepubescent children: the ExAMIN Youth South Africa study. J Hypertens. 2021 Nov 1;39(11):2190-2199. doi: 10.1097/HJH.0000000000002917. PMID 34620809
- [Derived] Kochli S, Botha-Le Roux S, Uys AS, Kruger R. Cardiorespiratory Fitness, Blood Pressure and Ethnicity Are Related to Salivary Cortisol Responses after an Exercise Test in Children: The ExAMIN Youth SA Study. Int J Environ Res Public Health. 2021 Jul 26;18(15):7898. doi: 10.3390/ijerph18157898. PMID 34360198
- [Derived] Kruger R, Monyeki MA, Schutte AE, Smith W, Mels CMC, Kruger HS, Pienaar AE, Gafane-Matemane LF, Breet Y, Lammertyn L, Mokwatsi GG, Kruger A, Deacon E, Hanssen H. The Exercise, Arterial Modulation and Nutrition in Youth South Africa Study (ExAMIN Youth SA). Front Pediatr. 2020 Apr 29;8:212. doi: 10.3389/fped.2020.00212. eCollection 2020. PMID 32411640
- See also: ORCID — https://orcid.org/0000-0001-7680-2032